CLINICAL TRIAL: NCT04284397
Title: Identification of Critical Thermal Environments for Aged Adults
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, W. Larry Kenney, Professor, Penn State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Study14062
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Aging
Keywords: Aging; Thermoregulation; Heat stress
MeSH Terms: conditions — Heat Stress Disorders | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Two groups of subjects (young, older) participate in twelve experiments; experimental conditions consist of six different combinations of temperature and humidity and are performed at two different exercise intensities. The experiments are conducted in randomized order and are separated by a minimum of three days. A subgroup of older adults will be asked to complete all trials after taking daily low-dose aspirin for seven days, and aspirin will be continued until all trials are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Critical Environmental Limits (Experimental): Subjects will perform exercise at ~200-300W with ambient temperature or humidity increasing every 5 min throughout the trial until core temperature begins to rise.
  Interventions: Other: Control
- Aspirin Supplementation (Experimental): After a minimum of 7 days of daily, low-dose aspirin ingestion, older subjects will repeat critical environmental limits trials. As before, subjects will perform exercise at ~200-300W with ambient temperature or humidity increasing every 5 min throughout the trial until core temperature begins to rise.
  Interventions: Drug: Low dose ASA

INTERVENTIONS:
Drug: Low dose ASA — A sub-group of older adults will be re-tested after 7 days of treatment with low-dose aspirin.
  Other Names: Low-dose aspirin
  Arms: Aspirin Supplementation
Other: Control — All participants will be tested with no treatment.
  Arms: Critical Environmental Limits

SUMMARY:
This study evaluates critical environmental limits (temperature and humidity) above which older adults are unable to effectively thermoregulate. Participants will exercise in a series of different environmental conditions to identify combinations of temperature and humidity above which age-related physiological changes cause uncompensable heat stress, resulting in increased risk of heat illness.

DETAILED DESCRIPTION:
The earth's climate is warming well above historical averages, and there is an increased frequency, duration, and severity of heat waves. At the same time, the world's population is rapidly aging. Aging is associated with reductions in thermoregulatory capacity due to reductions in sweating and skin blood flow. For this reason, people ≥65 years exhibit exponentially larger increases in morbidity and mortality during heat waves than younger individuals, with the large majority of excess deaths during heat waves occurring in the elderly.

Compounding the physiological effects of primary aging, co-morbidities and common classes of drugs taken by older adults can further compromise their thermoregulatory function. One such class of medications is cyclooxygenase inhibitors, including aspirin (ASA) and other platelet inhibitors. Provocative data published by our lab indicate that platelet inhibitors including ASA increase the rate of heat storage during passive heat stress by ~25%. Following current clinical guidelines, nearly 40% of US adults over the age of 50 engage in an aspirin therapy regiment for the primary or secondary prevention of cardiovascular disease.

Although there is compelling evidence that aging is associated with decreased heat dissipation and elevated risk of heat illness in hot ambient conditions, the significant question remains: In what specific environments does this age disparity begin to occur? The goal of the current study is to identify and model ambient conditions that are unsafe for older adults. A second aim of the study is to determine the effects of the commonly used platelet inhibitor, acetylsalicylic acid (ASA), on age-specific critical environmental limits.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older (those 40+ years of age must be cleared by collaborating physician)
* All premenopausal women will be eumenorrheic (by survey)
* Asymptomatic and no signs/symptoms of disease according to the American College of Sports Medicine 10th edition Guidelines for Exercise Testing and Prescription

Exclusion Criteria:

* Medications that affect thermoregulatory or cardiovascular responses to exercise
* Any contraindications to low intensity physical activity on the Physical Activity Readiness Questionnaire
* Any mobility restrictions that interfere with low intensity physical activity
* Pregnant or planning to become pregnant in the next 12 months
* Prior diagnosis of cancer, cardiovascular disease, diabetes, or metabolic syndrome
* Illegal/recreational drug use
* History of Chron's disease, diverticulitis, or similar gastrointestinal disease
* Abnormal resting or exercise electrocardiogram (ECG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2027-02-27 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
Temperature and humidity limits for maintaining stable core temperature | Through study completion, an average of 1 year.
  Core temperature will be measured throughout exercise. The point at which heat stress becomes uncompensable will be determined for each environmental and exercise condition by assessing the combination of temperature and humidity at which core temperature begins to rise.

SECONDARY OUTCOMES:
Core temperature | Continuous throughout visit until completion of exercise; an average of 2 hours.
  Core temperature will be monitored throughout each experimental visit
Sweat rate | Immediately before and immediately after exercise.
  Sweat rate will be determined by measuring nude body mass before and after each experimental visit
Skin temperature | Continuous throughout visit until completion of exercise; an average of 2 hours.
  Skin temperature will be monitored throughout each experimental visit

CONTACTS AND LOCATIONS:
Overall Officials: W. Larry Kenney, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No